CLINICAL TRIAL: NCT01815463
Title: Non-Invasive Prediction of Colorectal Neoplasia
Acronym: NIPCON
Status: Terminated | Type: Observational
Why Stopped: Local PI did not submit annual renewal, still active in Detroit, not recruiting.
Sponsor: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Martin Tobi, MB ChB, Corporal Michael J. Crescenz VA Medical Center
Other Study IDs: 00919; 0409000159 (Other Grant/Funding Number: 096294M1F)
Record Dates: First submitted 2013-03-18; First posted 2013-03-21 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Colonic Polyps; Polyposis Coli; Colorectal Cancer
Keywords: stool; monoclonal antibody; Adnab-9; FOBT; FIT; iFOBT; colonoscopy; barium enema; flexible sigmoidoscopy
MeSH Terms: conditions — Colonic Polyps; Adenomatous Polyposis Coli; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool Urine Saliva Blood Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- colorectal neoplasia: No interventions Record colorectal neoplasia

SUMMARY:
Hypothesis:The Adnab-9 antigen is a predictive biomarker in individuals at risk of developing colorectal neoplasia.

Study aim is to evaluate the potential of the Adnab-9 monoclonal antibody (MAb) as a marker of cancer risk in a population at increased risk for colorectal cancer (CRC). This marker would be compared to other current and emerging diagnostic methods. 2,800 Veterans would be recruited into the study. In phase 1, candidates would be defined as having increased CRC risk by a short questionnaire. Stool samples would be obtained and a semi-quantitative Adnab-9 antigen assay (ELISA) would be determined. Patients with differing high and low estimations of fecal Adnab-9 would undergo colonoscopy at which time other samples of effluent and colonic mucosa would be taken, and a detailed lifestyle and nutritional questionnaire would be completed. The characteristics of the Adnab-9 fecal test as a diagnostic test would be critically determined using the outcome of the colonoscopic and other test results. The patients will be contacted through the mail and by word of mouth. Informed consent will be obtained before the samples are obtained. The participants are clinically defined as high-risk and therefore screening colonoscopy would be likely performed in any event. A number of assays for Adnab-9 are feasible including slot-blot, Western blot, and ELISA. Other stool studies include conventional fecal occult blood tests (FOBT or FIT) that will be performed in tandem. The investigators therefore began this method of collection and obtained consent from over 2000 patients with a similar overall compliance rate with FOBT screening procedures to that reported previously of approximately 50%. Currently the study is no longer enrolling patients at the Detroit VA and is now finalizing data entry. Another 450 patients to be recruited at the Philadelphia VAMC.

DETAILED DESCRIPTION:
The primary objectives is to test the efficacy of Adnab-9 stool testing in a population at high-risk for colorectal neoplasia and directly compare it to that of the FOBT and secondarily, identify the source of the Adnab-9 antigen to determine influences of diet and environment on its expression. The design is a prospective cross sectional (Part 1) and a case-control longitudinal follow-up study (Part 2) using a brief questionnaire to assess risk for cancer in a total of 2800 Part I patients will be enrolled designed to achieve a database of high risk individuals and measure fecal Adnab-9 levels before a clinically indicated colonoscopy is performed. The patients submit 4 FOBT cards in a routine manner by mail, 3 are used for the FOBT and stool is extracted from the last card for the Adnab-9 ELISA which is reported as OD/5ug protein/well. 100 Part 2 enrollees are then selected on the basis of positive fecal Adnab-9 test candidates matched with a like number of patients with negative stool results who have had their initial colonoscopy and who will have a 5-year follow-up colonoscopy. Detailed Adnab-9 testing (immunohistochemical Adnab-9 binding; blood biomarker estimations and Adnab-9 Western blotting) will be performed on various bodily fluids to perfect the method of testing and completion of the detailed questionnaire to check for reproducibility and interim lifestyle changes in these participants.

ELIGIBILITY:
Inclusion Criteria:

* ability to complete a consent form
* must be at above average risk for colorectal neoplasia
* physically able to undergo colonoscopy or barium enema

Exclusion Criteria:

* Mentally handicapped
* Physically infirm
* Low risk for colorectal neoplasia
* Pregnant individuals
* Vulnerable populations

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Greater than average risk for colorectal neoplasia
Sampling Method: Probability Sample
Enrollment: 2282 (Actual)
Dates: Start 2006-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Correlation of Adnab-9 stool result with outcome of colonoscopy | 10 years
  Stool is collected on guaiac stool cards and/or stool Polymedco sample bottle and extracted. Extracted stool is assayed for protein content and this is used as a standard for the Adnab-9 ELISA. Record review note colonoscopy outcome which is correlated with Adnab-9 ELISA result.

SECONDARY OUTCOMES:
Define the origin of the Adnab-9 bound antigen | 10 years
  Biopsies are taken at the time of colonoscopy in ~10% of initial enrollees, from 6 colonic segments. In addition colonic effluent. saliva, urine and blood samples are taken. ELISA and immunohistochemistry for Adnab-9 binding are performed.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Tobi, MB,ChB, Principal Investigator — Philadelphia VAMC (WOC) Detroit VAMC (WOC) Saginaw VAMC; Fadi Antaki, MD, Principal Investigator — Detroit VAMC; John Lieb, MD, Principal Investigator — Philadelphia PVAMC
Locations (1):
- Philadelphia VAMC, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tobi M, Prabhu S, Gage RE, Orr T, Lawson MJ. Colorectal cancer risk: the impact of evidence of a field effect of carcinogenesis on blinded diagnosis using an anti-adenoma antibody test performed on colonoscopic effluent. Dig Dis Sci. 2002 Feb;47(2):317-21. doi: 10.1023/a:1013713920805. PMID 11855547
- [Background] Tobi M, Elitsur Y, Moyer MP, Halline A, Deutsch M, Nochomovitz L, Luk GD. Mucosal origin and shedding of an early colonic tumor marker defined by Adnab-9 monoclonal antibody. Scand J Gastroenterol. 1993 Dec;28(12):1025-34. doi: 10.3109/00365529309098304. PMID 8303203
- [Background] Tobi M, Maliakkal B, Zitron I, Alousi M, Goo R, Nochomovitz L, Luk G. Adenoma-derived antibody, Adnab-9 recognizes a membrane-bound glycoprotein in colonic tissue and effluent material from patients with colorectal neoplasia. Cancer Lett. 1992 Oct 30;67(1):61-9. doi: 10.1016/0304-3835(92)90009-k. PMID 1423246